CLINICAL TRIAL: NCT00937300
Title: T-cell Based Immunotherapy for Treatment of Patients Squamous Cell Carcinoma in the Oral Cavity. A Pilot Study.
Brief Title: T-cell Based Immunotherapy for Head and Neck Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The patients eligible for this trial do not exist anymore due to change in procedures.
Sponsor: Inge Marie Svane (Other)
Responsible Party: Sponsor-Investigator, Inge Marie Svane, Professor, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HH0908
Record Dates: First submitted 2009-07-10; First posted 2009-07-13 (Estimated); Last update posted 2011-11-23 (Estimated); Status verified 2011-11

CONDITIONS: Squamous Cell Carcinoma; Head and Neck Cancer
MeSH Terms: conditions — Carcinoma, Squamous Cell; Head and Neck Neoplasms | interventions — Cyclophosphamide; fludarabine; Interleukin-2; fludarabine phosphate; aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: cyclophosphamide, fludarabine, T-cell infusion, and Interleukin-2 — Two days of cyclophosphamide (60 mg/kg i.v.) and five days of fludarabine (25 mg/m2 i.v.). Infusion of Tumor Infiltrating Lymphocytes (10e9-10e10 cells). Followed by daily sc injections of 2 MIE Interleukin-2 for two weeks.
  Other Names: Cyclophosphamide, Sendoxan®, Baxter A/S; Fludarabine, Fludara®, Bayer Shering; Interleukin-2, Proleukin®, Chiron B.V.

SUMMARY:
The aim of this study is to investigate the toxicity and immune response of therapy with tumor infiltrating lymphocytes as adjuvant treatment for head and neck cancer after primary operation and radiotherapy.

Patient will receive a single treatment consisting of conditioning chemotherapy for seven days (cyclophosphamide for two days and fludarabine for five days), intravenous infusion of high number of in vitro expanded tumor infiltrating lymphocytes followed by two weeks with daily low-dose interleukine-2. Patients will be evaluated for toxicity and immune response.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histological proven squamous cell carcinoma T3 or more in the oral cavity planned for primary surgery. Performance Status 0 to 1. Acceptable CBC and blood chemistry results. Acceptable organ functions.

Exclusion Criteria:

* Patients with a history of any other malignancies less than five years ago. Brain metastases. Other significant illness including severe allergy, asthma, DM, angina pectoris, congestive heart failure, chronic infections, or active autoimmune disease. Treatment with immune suppressive drugs, experimental drugs, or antineoplastic drugs.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
toxicity | week 0 to 20

SECONDARY OUTCOMES:
immune response | week 0 to 20

CONTACTS AND LOCATIONS:
Overall Officials: Inge Marie Svane, Professor, MD, Study Director — Department of Oncology, Copenhagen University Hospital, Herlev, Herlev Ringvej 75, DK-2730 Herlev, Denmark
Locations (1):
- Department of Oncology, Copenhagen University Hospital, Herlev, Herlev, Denmark